CLINICAL TRIAL: NCT06528106
Title: Removal of Erroneous Penicillin Allergy Labels: Implementation Study (REPeAL)
Acronym: REPeAL
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2324.RCHT.66; 335337 (Other: IRAS); NIHR300542 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-06

CONDITIONS: Penicillin Allergy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To test the implementation of penicillin allergy de-labelling delivered by the responsible clinical teams and the antimicrobial stewardship teams across all medical, surgical and critical care specialities in a UK hospital using the developed toolkit and a validated penicillin allergy decision support tool.

DETAILED DESCRIPTION:
Aim:

To test implementation of the penicillin allergy de-labelling complex intervention in surgical, medical and critical care patient pathway.

Objectives:

* To use the Institute for Health Improvement (IHI) Model for Improvement methodology to implement the penicillin allergy de-labelling complex intervention in each setting (surgery, medicine, critical care)
* To measure the number of patients meeting inclusion criteria (>16 with a penA not prescribed first line antibiotics) who have had their penicillin allergy record assessed by the wider clinical teams and separately by the AMS team.
* To measure the patient uptake of penicillin allergy record removal (i.e. the rate of patient declining de-label / DOC).

To interview 10-15 patients and 10-15 healthcare workers to gain insight into the penicillin allergy de labelling process.

ELIGIBILITY:
Inclusion Criteria:

All adult (>16) patients admitted to hospital over the study period with a penicillin allergy record preventing first line antibiotic use.

Exclusion Criteria:

None

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult (>16) patients admitted to hospital over the study period with a penicillin allergy record preventing first line antibiotic use.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients admitted to adult medical, surgical and critical care specialities with a penicillin allergy record, where the allergy record is preventing first line antibiotic therapy, that are safely de-labelled. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No